CLINICAL TRIAL: NCT03420599
Title: Altered Microbiota is Related Increased Infection Rates After Traumatic Splenectomy
Brief Title: Microbiota is Related With Increasing Infection Rates After Splenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2017-12-20
Record Dates: First submitted 2017-12-24; First posted 2018-02-05 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-12

CONDITIONS: Gut Microbiota; Spleen Injury; Infection
Keywords: Gut microbiota; Splenectomy; Infection; Immune; Cytokines
MeSH Terms: conditions — Infections | interventions — Splenectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- health control: healthy controls are all from normal volunteers
- splenectomy: Traumatic patients after total splenectomy
  Interventions: Procedure: splenectomy

INTERVENTIONS:
Procedure: splenectomy — Traumatic patients who performed total splenectomy
  Groups: splenectomy

SUMMARY:
Studies has shown an increasingly infection rate after splenectomy, and there is a potential correlation between microbiota and immune system. investigators suppose that increasingly infection can be associated with the alteration composition of the gut microbiota after splenectomy. It's investigators' aim to discover if any difference of gut microbiota is exist in patients who suffer from traumatic splenectomy compared with normal people, ultimately aim toreduce and mitigation infection rate through controlling gut microbiota.

DETAILED DESCRIPTION:
The spleen is crucial in regulating immune homoeostasis through its ability to link innate and adaptive immunity and to protect against infections. Asplenia refers to the absence of the spleen, a disorder that is rarely congenital and is more frequently as a result of surgery. Splenic hypofunction, as a result of asplenia can lead a series of changes in body systems. Recent study has show an increasingly infection rate after splenectomy including abdominal infection, pulmonary infection and cranial cavity infection.

The gastrointestinal tract plays host to a diverse and metabolically complex community of microorganisms. Recent literature suggests that organisms in the gastrointestinal tract, referred to collectively as gut microbiota, play an indispensable role in the maintenance of host's homeostasis. Study has proved a potential correlation between microbiota and immune system. Lymphocyte, in either peripheral circulation or mesenteric lymph node, altered can lead to an composition change in microbiota.

Investigators suppose that this phenomenon can be associated with the alteration of the resident commensal microenvironment after splenectomy compared to commensal communities. It's investigators' aim to discover if any difference of gut microbiota is exist in patients who suffer from traumatic splenectomy compared with normal people, ultimately aim toreduce and mitigation infection rate through controlling gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* All the patients underwent an total splenectomy in the First Affiliated Hospital of Harbin Medical University from January 1st, 2015 to May 1st, 2017. Each participant provided a fresh stool sample in hospital when following-up.

Exclusion Criteria:

* Use antibiotics and probiotics 3 mouth before samples collection.
* Other severe abdomen injury
* Underwent abdomen organ resection surgery
* Other digestive system disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population are aged from 18 to 65 years，which divided into 2 groups: Splenectomy, healthy controls
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-11-25 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
Transcriptional changes in gut microbiota | Baseline, 6 months after surgery, 12 months after surgery, 24 months after surgery
  16S rRNA gene sequencing will be performed with stander procedure
Transcriptional changes in plasma LPS levels | Baseline, 6 months after surgery, 12 months after surgery, 24 months after surgery
  Plasma LPS level will be measured by ELISA

SECONDARY OUTCOMES:
Fecal SIgA | Baseline, 6 months after surgery, 12 months after surgery, 24 months after surgery
  Fecal SIgA antibody will be measured by ELISA
Fecal calprotectin | Baseline, 6 months after surgery, 12 months after surgery, 24 months after surgery
  Fecal SIgA antibody will be measured by ELISA
Plasma DAO | Baseline, 6 months after surgery, 12 months after surgery, 24 months after surgery
  Plasma DAO antibody will be measured by ELISA
Plasma D-Lac | Baseline, 6 months after surgery, 12 months after surgery, 24 months after surgery
  Plasma D-Lac antibody will be measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yunwei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China